CLINICAL TRIAL: NCT05420259
Title: Influence of a Combined Dietary and Exercise Intervention on Cytokine Profile and NK Cell Activation in Cancer Patients Undergoing Neoadjuvant Treatment.
Brief Title: Combined Exercise and Nutritional Intervention in GI Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Beatriz Ângelo (Other)
Responsible Party: Principal Investigator, Sónia Velho, Nutricionist, Hospital Beatriz Ângelo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 213/18
Record Dates: First submitted 2022-06-13; First posted 2022-06-15 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Pancreatic Cancer; Gastric Cancer; Diet; Exercise
Keywords: Body composition; Wasting; Malnutrition
MeSH Terms: conditions — Pancreatic Neoplasms; Stomach Neoplasms; Motor Activity; Cachexia; Malnutrition | interventions — Diet Therapy; Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined Exercise and Dietary Intervention (Experimental): Intervention aimed at conveying a supervised combined moderate aerobic and resistance training, once a week with a duration of 40-60 minutes plus daily home exercise, personalized according to patients' age and functional status. Dietary intervention aimed at a one-on-one nutritional counseling. In the first visit a dietary plan is designed and one daily oral nutritional supplement (Fortimel Compact®, Nutricia) is given to meet the European Society of Parenteral and Enteral Nutrition (ESPEN) recommended intake.
  Interventions: Behavioral: Combined Exercise and Dietary Intervention (CEDI)
- Control (Other): Standard Care
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Combined Exercise and Dietary Intervention (CEDI) — The exercise program will be planned by an exercise physiologist and implemented by physiotherapists prior to rehabilitation physician assessment. In the first session patients will be evaluated by physiotherapist in order to allow personalization of exercise according to patient's age and functional capacity. In regard to diet, written materials will be given to patients and caregivers, namely a dietary plan, standard menus, recipes, and standard portions information.
  Arms: Combined Exercise and Dietary Intervention
Behavioral: Standard Care — Standard Care
  Arms: Control

SUMMARY:
Although some studies have focused on the role of exercise on inflammation and cytokine expression in cancer patients undergoing treatment and survivors, to our knowledge none have investigated the effect of exercise during neoadjuvant treatment as a complementary therapy to 1) modulate inflammation which may have a positive influence on chemotherapy response and 2) preserve or improve skeletal muscle, thus preventing cancer cachexia. Furthermore, we believe that the neoadjuvant treatment period could be a window of opportunity to optimize patient's nutritional status before surgery, which until now has been under used.

Bearing in mind that nutritional interventions may also influence IL-6, our hypothesis is that a Combined Exercise and Dietary Intervention (CEDI) may induce positive alterations in cytokine profile and increase NK cell infiltration of the tumor in gastric and pancreatic cancer patients submitted to neo-adjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* gastric or pancreatic cancer stage II/III, eligible for neoadjuvant chemotherapy,
* age higher than 40 years and lower than 80 years,
* ECOG (Eastern Cooperative Oncology Group) functional status: 0-2,
* sedentary/low physical activity level.

Exclusion Criteria:

* life expectancy less than 12 months at inclusion,
* chemotherapy regimen other than 5-Fluorouracil, Folinic acid, Oxaliplatin, Docetaxel (FLOT) for gastric and 5-Fluorouracil, Irinotecan and Oxaliplatin (FOLFIRINOX) or gemcitabine for pancreatic cancer,
* metastatic disease,
* chronic anti-inflammatory medication use,
* known inflammatory condition (rheumatoid arthritis, ankylosing spondylitis or chronic active hepatitis)
* cardiovascular, respiratory or musculoskeletal or joint problems that preclude moderate physical activity.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2024-06-28 (Estimated); Study Completion 2024-06-28 (Estimated)

PRIMARY OUTCOMES:
Mean Change in interleukin 6 (IL6) | 8 weeks
  IL6 circulating levels will be determined before and after combined exercise and dietary intervention (CEDI)

SECONDARY OUTCOMES:
Change in Immune cell infiltration profile on tumor specimen | 8 weeks
  Peri-tumoral cell distribution (NK cells, T cells) will be determined before and after combined exercise and dietary intervention (CEDI)
Change in skeletal muscle | 8 weeks
  Skeletal muscle using CT scan body composition analysis will be assessed before and after combined exercise and dietary intervention (CEDI)

CONTACTS AND LOCATIONS:
Overall Officials: Marilia Cravo, Study Director — Hospital da Luz
Locations (2):
- Portugal (2):
  - Hospital Beatriz Ângelo, Loures, Lisbon District
  - Hospital da Luz, Lisbon

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP